CLINICAL TRIAL: NCT02193776
Title: A Phase 2 Open-Label Partially Randomized Trial to Evaluate the Efficacy, Safety and Tolerability of Combinations of Bedaquiline, Moxifloxacin, PA-824 and Pyrazinamide During 8 Weeks of Treatment in Adult Subjects With Newly Diagnosed Drug-Sensitive or Multi Drug-Resistant, Smear-Positive Pulmonary Tuberculosis.
Brief Title: A Phase 2 to Evaluate the Efficacy, Safety and Tolerability of Combinations of Bedaquiline, Moxifloxacin, PA-824 and Pyrazinamide in Adult Subjects With Drug-Sensitive or Multi Drug-Resistant Pulmonary Tuberculosis.
Acronym: NC-005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC-005-(J-M-Pa-Z)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Multi Drug-Resistant Tuberculosis; Drug-Sensitive Tuberculosis; PA-824; Bedaquiline; Moxifloxacin; Pyrazinamide; Quinolone; Pretomanid; NC-005
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — pretomanid; bedaquiline; Moxifloxacin; Pyrazinamide; Isoniazid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DS-TB: J(loading dose/t.i.w.)PaZ (Experimental): Subjects with DS-TB. J(loading dose/t.i.w.)PaZ: Bedaquiline 400mg once daily Days 1-14, 200mg three times per week Days 15-56; plus PA-824 200mg once daily Days 1-56; plus pyrazinamide 1500mg once daily Days 1-56.
  Interventions: Drug: PA-824; Drug: bedaquiline; Drug: pyrazinamide
- DS-TB: J(200mg)PaZ (Experimental): Subjects with DS-TB. J(200mg)PaZ: Bedaquiline 200mg once daily Days 1-56; plus PA-824 200mg once daily Days 1-56; plus pyrazinamide 1500mg once daily Days 1-56.
  Interventions: Drug: PA-824; Drug: bedaquiline; Drug: pyrazinamide
- MDR-TB: J(200mg)MPaZ (Experimental): Subjects with MDR-TB. J(200mg)MPaZ: Bedaquiline 200mg once daily Days 1-56; plus moxifloxacin 400mg once daily Days 1-56; plus PA-824 200mg once daily Days 1-56; plus pyrazinamide 1500mg once daily Days 1-56.
  Interventions: Drug: PA-824; Drug: bedaquiline; Drug: moxifloxacin; Drug: pyrazinamide
- DS-TB: HRZE (Active Comparator): Subjects with DS-TB. HRZE tablets (Isoniazid 75mg plus rifampicin 150mg plus pyrazinamide 400mg plus ethambutol 275mg combination tablets) dosed once daily Days 1-56 per the Subject's weight as follows: 30-37kg: 2 tablets; 38-54kg: 3 tablets; 55-70kg: 4 tablets; 71kg and over: 5 tablets.
  Interventions: Drug: isoniazid, rifampicin, pyrazinamide and ethambutol combination tablet

INTERVENTIONS:
Drug: PA-824 — oral
  Arms: DS-TB: J(200mg)PaZ; DS-TB: J(loading dose/t.i.w.)PaZ; MDR-TB: J(200mg)MPaZ
Drug: bedaquiline — oral
  Other Names: TMC207; Sirturo
  Arms: DS-TB: J(200mg)PaZ; DS-TB: J(loading dose/t.i.w.)PaZ; MDR-TB: J(200mg)MPaZ
Drug: moxifloxacin — oral
  Other Names: BAY 12-8039; Avelox; Avalon; Avelon
  Arms: MDR-TB: J(200mg)MPaZ
Drug: pyrazinamide — oral
  Arms: DS-TB: J(200mg)PaZ; DS-TB: J(loading dose/t.i.w.)PaZ; MDR-TB: J(200mg)MPaZ
Drug: isoniazid, rifampicin, pyrazinamide and ethambutol combination tablet — oral
  Arms: DS-TB: HRZE

SUMMARY:
The purpose of this study is to determine the mycobactericidal activity of combinations of bedaquiline (J), moxifloxacin (M), PA-824 (Pa) and pyrazinamide (Z) regimens during 8 weeks of treatment.

DETAILED DESCRIPTION:
The trial design is a phase 2, multi-center, open-label, partially randomized clinical trial in four parallel treatment groups. Subjects with drug-sensitive tuberculosis (DS-TB) will be randomized to receive either J(loading dose/three times a week)PaZ; or J(200mg)PaZ; or HRZE. Subjects with multi drug-resistant tuberculosis will receive J(200mg)MPaZ. The HRZE treatment arm is included as a control for the drug-sensitive treatments and as a control for the quantitative laboratory mycobacteriology testing.

A total of approximately 240 male and female, newly diagnosed subjects with drug-sensitive or multi drug-resistant, smear positive pulmonary tuberculosis aged 18 to 75 years (inclusive) will be included in the study. A total of 180 subjects with drug-sensitive tuberculosis (60 per treatment arm) will be randomized. Up to 60 subjects with multi-drug resistant tuberculosis will be assigned.

All subjects will have up to a maximum of 9 days screening, receive 8 weeks of treatment, and have follow-up visits at 2 and 12 weeks after study treatment completion or last dose of investigational medicinal product in the case of early withdrawal. Subjects who withdraw from the study after receiving < 14 days of investigational medicinal product, will only attend a follow-up visit at 2 weeks after last dose of investigational medicinal product.

Upon treatment completion, the subjects with drug-sensitive tuberculosis will be provided with sufficient doses of standard of care tuberculosis treatment, as appropriate, to cover the time period from attending their last visit at the study clinic until their scheduled visit at the TB clinic. All subjects with drug sensitive and multi-drug resistant tuberculosis will be referred to the local community tuberculosis clinics for standard anti-tuberculosis chemotherapy according to National Tuberculosis Guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures. Male or female, aged between 18 and 75 years inclusive.
2. Body weight (in light clothing and with no shoes) between 35 and 100 kg, inclusive.
3. Tested at the trial appointed laboratory: M. Tb positive on molecular test (e.g. GeneXpert or Hain) and sputum smear-positive pulmonary TB on direct microscopy for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale.

   * For DS-TB treatment arms (defined as sensitive to rifampicin based on molecular sensitivity testing), Subjects should be:

     1. either newly diagnosed or untreated for at least 3 years after cure from a previous episode (Subject can give a history of cure and previous treatment); AND
     2. Previous TB treatment must be discontinued as per exclusion criteria 16.
   * For MDR-TB treatment arm (defined as resistant to rifampicin based on molecular sensitivity testing), Subjects should be:

     1. sensitive to moxifloxacin by molecular sensitivity testing; AND
     2. either newly diagnosed or could have previously been treated for DS-TB and/or MDR-TB (< 7 days of treatment). Previous MDR-TB treatment must be discontinued as per exclusion criteria 17.
4. A chest X-ray picture which in the opinion of the Investigator is compatible with TB.
5. Ability to produce an adequate volume of sputum as estimated from a screening Coached Spot Sputum Sample assessment (estimated 10 ml or more overnight production).
6. Be of non-childbearing potential or using effective methods of birth control, as defined below:

Non-childbearing potential:

1. Subject - not heterosexually active or practices sexual abstinence; or
2. Female Subject/sexual partner - bilateral oophorectomy, bilateral tubal ligation and/or hysterectomy or has been postmenopausal with a history of no menses for at least 12 consecutive months; or
3. Male Subject/sexual partner - vasectomised or has had a bilateral orchidectomy minimally three months prior to screening.

Effective birth control methods:

A double contraceptive method should be used as follows:

1. Double barrier method which can include any 2 of the following: a male condom, diaphragm, cervical cap, or female condom (male and female condoms should not be used together); or
2. Barrier method (one of the above) combined with hormone-based contraceptives or an intra-uterine device for the female Subject/partner; and are willing to continue practicing birth control methods throughout treatment and for 6 months (both male and female Subjects) after the last dose of study medication or discontinuation from study medication in case of premature discontinuation.

(Note: Hormone-based contraception alone may not be reliable when taking IMP; therefore, hormone-based contraceptives alone cannot be used by female Subjects or female partners of male Subjects to prevent pregnancy).

Exclusion Criteria:

Medical Criteria

1. Evidence of clinically significant (as judged by the Investigator), metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied) including malaria. A rapid test for malaria may be carried out if indicated.
2. Karnofsky performance status score of < 60%.
3. Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
4. Clinically significant evidence of extrathoracic TB (e.g. miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
5. History of allergy or hypersensitivity to any of the study Investigational Medicinal Products or related substances.
6. Known or suspected current alcohol and/or drug abuse (positive urine drug screen) or history thereof within the past 2 years that is, in the opinion of the Investigator, sufficient to compromise the safety and/or cooperation of the Subject.
7. For HIV infected Subjects:

   1. having a CD4+ count <100 cells/µL;
   2. with an AIDS-defining opportunistic infection or malignancies (except pulmonary TB);
   3. currently treated with or will need to initiate antiretroviral therapy (ART) which is not compatible with the allowed ARTs and is not considered an appropriate candidate for switching to a regimen of ARVs which is allowed as follows:

      * Triple nucleoside reverse transcriptase inhibitor (NRTI) based regimen consisting of zidovudine, lamivudine, and abacavir;
      * Nevirapine based regimen consisting of nevirapine in combination with any NRTIs;
      * Lopinavir/ritonavir (Aluvia™) based regimen consisting of lopinavir/ritonavir (Aluvia™) in combination with any NRTIs;
      * Raltegravir in combination with nucleoside reverse transcriptase inhibitors (NRTIs);
   4. cannot ensure a 2 week interval between commencing IMP and the start of ART.
8. Having participated in other clinical study/ies with investigational agent/s within 8 weeks prior to trial start.
9. Significant cardiac arrhythmia requiring medication.
10. Subjects with the following at screening (per measurements and reading done by Central ECG):

    1. Marked prolongation of QT/QTc interval, e.g. confirmed demonstration of QTcF (Fridericia correction) or QTcB (Bazett correction) interval >450 ms at screening;
    2. History of additional risk factors for Torsade de Pointes, e.g. heart failure, hypokalemia, family history of Long QT Syndrome;
    3. Use of concomitant medications that are known to prolong the QT/QTc interval (see exclusion criteria 19);
    4. Any clinically significant, in the opinion of the Investigator, ECG abnormality.
11. Females who are pregnant, breast-feeding, or planning to conceive a child during the study or within 6 months of cessation of treatment. Males planning to conceive a child during the study or within 6 months of cessation of treatment.
12. Diabetes Mellitus resulting in hospitalization in the past year.
13. Evidence of lens opacity on slit lamp ophthalmologic examination as defined by a grading of >1+ on the AREDS2 grading system.
14. For males, any history of a clinically significant abnormality in the reproductive system.

    Specific Treatments
15. Previously received treatment with PA-824, bedaquiline or moxifloxacin as part of a clinical trial.
16. For the DS-TB treatment arms: treatment with any drug active against M. Tb within the 3 years prior to Day 1 (including but not limited to isoniazid, ethambutol, amikacin, bedaquiline, clofazimine, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides, metronidazole). Exceptions include the use of fluoroquinolones and metronidazole as short-term treatment (≤2 weeks) for Non-M.Tb infections. Treatment should have been discontinued at least 3 months prior to Day 1. Subjects who have previously received isoniazid prophylactically may be included in the trial as long as that treatment is/was discontinued at least 7 days prior to randomization into this trial.
17. MDR-TB Subjects may have previously been treated for DS-TB with first-line TB drugs (isoniazid, rifampicin, ethambutol, pyrazinamide and/or streptomycin) and/or received ≤7 days MDR-TB treatment, provided that treatment is/was discontinued at least 7 days prior to randomization. It should be confirmed that the MDR-TB treatment can be safely stopped and the screening period is long enough to allow for a washout period of 5 times the longest half-life of the drugs.
18. Any diseases or conditions in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to acute gout, allergy to any TB drug, their component or to the IMP.
19. Use of any drug within 30 days prior to dosing known to prolong QTc interval (including but not limited to amiodarone, bepridil, chloroquine, chlorpromazine, cisapride, cyclobenzaprine, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, thioridazine). Exceptions may be made for Subjects that have received 3 days or less of one of these drugs or substances, if there has been a wash-out period before administration of IMP equivalent to at least 5 half-lives of that drug or substance. Subjects who have taken drugs with long elimination half-lives such as amiodarone should be discussed with the Sponsor.
20. Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes (including but not limited to quinidine, tyramine, ketoconazole, fluconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan). Exceptions may be made for Subjects that have received 3 days or less of one of these drugs or substances, if there has been a wash-out period before administration of IMP equivalent to at least 5 half-lives of that drug or substance.
21. Any ARVs other than allowable ARVs detailed in exclusion criteria no. 7 above.

    Based on Laboratory Abnormalities:
22. Subjects with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table:

    1. serum magnesium and calcium (corrected for albumin) levels outside of the laboratory's reference range
    2. lipase grade 3 or greater (>2.0 x ULN);
    3. creatinine grade 2 or greater (>1.5 x ULN);
    4. hemoglobin grade 4 (<6.5 g/dL);
    5. platelets > grade 2 (under 50x10(9) cells/L);
    6. serum potassium less than the lower limit of normal for the laboratory;
    7. aspartate aminotransferase (AST) grade 3 or greater (≥3.0 x ULN) to be excluded;
    8. alanine aminotransferase (ALT) grade 3 or greater (≥3.0 x ULN) to be excluded;
    9. alkaline phosphatase (ALP) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 - 8.0 x ULN) must be discussed with and approved by the Sponsor Medical Monitor;
    10. total bilirubin grade 3 or greater (≥2.0 x ULN, or ≥1.50 x ULN when accompanied by any increase in other liver function test) to be excluded, grade 2 (≥1.50 x ULN, or ≥1.25 x ULN when accompanied by any increase in other liver function test) must be discussed with and approved by the Sponsor Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2016-02-08 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Dawson, Principal Investigator — University of Cape Town Lung Institute
Locations (10):
- South Africa (7):
  - The Aurum Institute: Tembisa Hospital, Tembisa, Gauteng
  - Klerksdorp Tshepong Hospital, Jouberton, Klerksdorp
  - TASK Applied Science, Cape Town
  - University of Cape Town Lung Institute (Pty) Ltd, Cape Town
  - THINK: Tuberculosis & HIV Investigative Network of KwaZulu-Natal, Durban
  - CHRU Themba Lethu Clinic, Johannesburg
  - University of Witwatersrand, Clinical HIV Research Unit (CHRU), Helen Joseph Hospital, Johannesburg
- Tanzania (2):
  - Ifakara Health Institute, Bagamoyo
  - NIMR-Mbeya Medical Research Centre (MMRC), Mbeya
- Uganda Case Western Reserve University Research Collaboration, Kampala, Uganda

REFERENCES:
- [Derived] Tweed CD, Dawson R, Burger DA, Conradie A, Crook AM, Mendel CM, Conradie F, Diacon AH, Ntinginya NE, Everitt DE, Haraka F, Li M, van Niekerk CH, Okwera A, Rassool MS, Reither K, Sebe MA, Staples S, Variava E, Spigelman M. Bedaquiline, moxifloxacin, pretomanid, and pyrazinamide during the first 8 weeks of treatment of patients with drug-susceptible or drug-resistant pulmonary tuberculosis: a multicentre, open-label, partially randomised, phase 2b trial. Lancet Respir Med. 2019 Dec;7(12):1048-1058. doi: 10.1016/S2213-2600(19)30366-2. Epub 2019 Nov 12. PMID 31732485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 10 centers in 3 countries (South Africa, Tanzania, and Uganda) from 23 October 2014. Adult male and female participants with drug-sensitive (DS) or multi-drug resistant (MDR) smear-positive pulmonary tuberculosis (TB) were recruited into this open-label multi-center study.
Pre-assignment Details: Participants were confirmed positive for M.tuberculosis on molecular test. DS-TB participants were to be sensitive to rifampicin and newly diagnosed with pulmonary TB (or untreated for at least 3 years). MDR-TB participants were to be resistant to rifampicin, sensitive to moxifloxacin and newly diagnosed with pulmonary TB (or treated for <=7 days).
Groups:
- DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide: Participants with DS-TB were randomized to receive 400 milligrams (mg) bedaquiline once daily on Days 1 to 14, 200 mg three times a week (t.i.w) during Days 15 to 56 + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily on Days 1 to 56 during the treatment period (from Day 1 to Week 8). Participants then entered a follow-up period up to Month 26.
- DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide: Participants with DS-TB were randomized to receive 200 mg bedaquiline + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily on Days 1 to 56 during the treatment period (from Day 1 to Week 8). Participants then entered a follow-up period up to Month 26.
- DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol): Participants with DS-TB were randomized to receive combination tablets containing 75 mg isoniazid + 150 mg rifampicin + 400 mg pyrazinamide + 275 mg ethambutol orally once daily on Days 1 to 56 during the treatment period (from Day 1 to Week 8) with the daily dose per the participant's weight as follows: 30 to 37 kilograms (kg): 2 tablets; 38 to 54 kg: 3 tablets; 55 to 70 kg: 4 tablets; 71 kg and over: 5 tablets. Participants then entered a follow-up period up to Month 26.
- MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide: Participants with MDR-TB received 200 mg bedaquiline + 400 mg moxifloxacin + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily on Days 1 to 56 during the treatment period (from Day 1 to Week 8). Participants then entered a follow-up period up to Month 26.
Period: Overall Study
Arm/Group | DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide | DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide | DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol) | MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide
Started | 59 | 60 | 61 | 60
Completed Day 70 Follow-up | 54 | 56 | 60 | 60
Completed Day 140 Follow-up | 52 | 52 | 58 | 58
Completed (Completed Treatment) | 51 | 53 | 59 | 58
Not Completed | 8 | 7 | 2 | 2
Not completed — Consent withdrawn | 1 | 0 | 0 | 0
Not completed — Failure to comply with protocol | 0 | 1 | 0 | 0
Not completed — Investigator/Sponsor decision | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse event/Specific toxicity | 5 | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis population included all participants who were randomized (for the DS participant population) or assigned (for the MDR participant population) to study drug and who received at least 1 administration of study drug.
Groups:
- DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide: Participants with DS-TB were randomized to receive 400 mg bedaquiline once daily on Days 1 to 14, 200 mg t.i.w during Days 15 to 56 + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily on Days 1 to 56 during the treatment period (from Day 1 to Week 8). Participants then entered a follow-up period up to Month 26.
- DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol): Participants with DS-TB were randomized to receive combination tablets containing 75 mg isoniazid + 150 mg rifampicin + 400 mg pyrazinamide + 275 mg ethambutol orally once daily on Days 1 to 56 during the treatment period (from Day 1 to Week 8) with the daily dose per the participant's weight as follows: 30 to 37 kg: 2 tablets; 38 to 54 kg: 3 tablets; 55 to 70 kg: 4 tablets; 71 kg and over: 5 tablets. Participants then entered a follow-up period up to Month 26.
- Total: Total of all reporting groups
Arm/Group | DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide | DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide | DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol) | MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide | Total
Number analyzed (Participants) | 59 | 60 | 61 | 60 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (13.03) | 33.9 (10.45) | 33.3 (8.60) | 34.0 (12.68) | 34.1 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 15 | 17 | 58
  Male | 45 | 48 | 46 | 43 | 182
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 46 | 49 | 49 | 53 | 197
  White | 0 | 0 | 0 | 1 | 1
  More than one race | 13 | 11 | 12 | 5 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Time to Sputum Culture Positivity (TTP) Over 8 Weeks in the Mycobacterial Growth Indicator Tube (MGIT) System
Description: The bactericidal activity (BA) was determined by the rate of change in TTP collected from overnight sputum samples over 8 weeks of treatment in the liquid culture media MGIT system, represented by the model-fitted log(TTP) results as calculated by the regression of the observed log(TTP) results over time. The bactericidal activity of log(TTP) over Day 0 to Day 56 (BATTP[0-56]) was presented and expressed as the daily percentage change in TTP from Day 0 to Day 56. The mean BATTP (0-56) was calculated from Bayesian non-linear mixed effects regression models fitted to log(TTP) collected from sputum samples (observed from Day 0 to Day 56).
Time Frame: Day 0 to Day 56 (8 weeks)
Population: The modified intention-to-treat analysis population included all participants included in the safety analysis population for whom valid corresponding efficacy data were available. Pyrazinamide resistant participants were excluded from this analysis population (applicable to both participants with DS-TB and MDR-TB).
Measure: Mean (Standard Deviation); unit: percentage change in TTP/day
Arm/Group | DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide | DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide | DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol) | MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide
Number analyzed (Participants) | 57 | 56 | 59 | 37
percentage change in TTP/day | 4.878 (1.604) | 5.182 (1.466) | 4.046 (1.129) | 5.194 (1.068)

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any AE which started or worsened on or after first study drug administration up to and including the Day 70 follow-up visit (or up to and including 14 days after last study drug administration for participants not having Day 70 follow-up visit). Drug-related TEAEs were defined as TEAEs for which relationship to study drug was indicated as 'possible', 'probable', 'certain' or missing. TEAEs leading to death were defined as TEAEs resulted 'fatal' outcome. Serious TEAEs were defined as TEAEs for which serious was indicated as 'yes'. TEAEs leading to discontinuation of study drug were defined as TEAEs for which action taken with study drug was indicated as 'study drug stopped'. TEAEs leading to early withdrawal from study were defined as TEAEs resulted study discontinuation. Grade III and IV TEAEs were defined as TEAEs for which severity (DMID grade) was indicated as 'Grade 3 (severe)' and 'Grade 4 (potentially life-threatening)' or missing, respectively.
Time Frame: First study drug administration (Day 1) up to and including the Day 70 follow-up visit (or up to and including 14 days after last study drug administration for participants not having the Day 70 follow-up visit) (70 days)
Population: The safety analysis population included all participants who were randomized (for the DS participant population) or assigned (for the MDR participant population) to study drug and received at least 1 administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide | DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide | DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol) | MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide
Number analyzed (Participants) | 59 | 60 | 61 | 60
Participants
  Any TEAE | 50 | 45 | 44 | 57
  Drug-related TEAE | 38 | 29 | 29 | 46
  TEAE leading to death | 1 | 1 | 1 | 0
  Any serious TEAE | 4 | 3 | 4 | 4
  Drug-related serious TEAE | 2 | 0 | 1 | 2
  TEAE leading to discontinuation of study drug | 6 | 5 | 2 | 2
  TEAE leading to early withdrawal from study | 5 | 5 | 2 | 2
  Grade III TEAE | 19 | 17 | 14 | 13
  Grade IV TEAE | 8 | 7 | 2 | 1

ADVERSE EVENTS:
Time Frame: TEAEs were collected from first study drug administration (Day 1) up to and including the Day 70 follow-up visit (or up to and including 14 days after last study drug administration for participants not having the Day 70 follow-up visit) (70 days).
Description: The safety analysis population included all participants who were randomized (for the DS participant population) or assigned (for the MDR participant population) to study drug and received at least 1 administration of study drug. All-cause mortality is defined as death due to any cause for entire duration of study.
Arm/Group | DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide | DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide | DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol) | MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide
All-Cause Mortality (participants affected / at risk) | 2/59 | 3/60 | 2/61 | 4/60
Serious Adverse Events (participants affected / at risk) | 4/59 | 3/60 | 4/61 | 4/60
Other Adverse Events (participants affected / at risk) | 50/59 | 45/60 | 44/61 | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide (N=59) | DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide (N=60) | DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol) (N=61) | MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide (N=60)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Malaria (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-TB: Bedaquiline (Loading Dose/t.i.w)+ PA-824 + Pyrazinamide (N=59) | DS-TB: Bedaquiline (200 mg) + PA-824 + Pyrazinamide (N=60) | DS-TB: HRZE (Isoniazid+Rifampicin+Pyrazinamide+Ethambutol) (N=61) | MDR-TB: Bedaquiline (200 mg)+Moxifloxacin+PA-824+Pyrazinamide (N=60)
Blood uric acid increased (Investigations) | 15 | 13 | 9 | 27
Alanine aminotransferase increased (Investigations) | 3 | 5 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 3 | 3
Amylase increased (Investigations) | 0 | 0 | 1 | 10
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 5 | 6 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 4
Influenza (Infections and infestations) | 3 | 0 | 3 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 4
Vomiting (Gastrointestinal disorders) | 4 | 1 | 4 | 7
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6 | 6
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 | 4 | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator or any Sub-Investigator shall submit any oral or written publication or abstract concerning this study to the Sponsor not less than thirty (30) days prior to submission to any journal, other publication or meeting for review and removal of confidential information.

DOCUMENTS (2):
  • Study Protocol (2014-09-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT02193776/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02193776/SAP_001.pdf